CLINICAL TRIAL: NCT03800823
Title: A Randomized Controlled Trial for Overweight and Obesity in Preschoolers - The More and Less Study Europe
Brief Title: Overweight and Obesity in Preschoolers
Acronym: MLEurope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other); El Centro de Investigación Biomédica en Red, CIBER (Unknown)
Responsible Party: Principal Investigator, Paulina Nowicka, Senior Researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 774548-WP8
Record Dates: First submitted 2019-01-02; First posted 2019-01-11 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Overweight
Keywords: Children; Obesity; Treatment; Family; mHealth
MeSH Terms: conditions — Obesity; Overweight | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent group & mHealth component (Experimental): The intervention in the present study is a 10 week parent training group session (More and Less Program) followed by a 6-month mobile phone based intervention. Both components aim to develop healthy lifestyle behaviours regarding dietary habits and physical activity in 2-6 year olds. The intervention is delivered towards the parents.
  Interventions: Behavioral: Parent group; Behavioral: mHealth component
- Standard care (Active Comparator): Standard care for overweight and obesity
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Parent group — In group sessions parents will learn how to use positive parenting practices (e.g., encouragement and limit setting) instead of ineffective practices (e.g., coercive behaviour, negative reciprocity). Using a parent group approach, each of the 10 sessions consist of introduction to effective parenting practices followed by a discussion and practice using role play and home practice assignments.
  Arms: Parent group & mHealth component
Behavioral: mHealth component — After the group sessions, parents will receive a 6-month mHealth program (MINISTOP app) based on social cognitive theory with strategies to change unhealthy diet/physical activity behaviours. The program includes information, advice, and strategies to change unhealthy behaviours and the possibility to register the child's intake of fruit, vegetables, candy, sweetened beverages, and sedentary time.
  Arms: Parent group & mHealth component
Behavioral: Standard care — Standard care for overweight and obesity.
  Arms: Standard care

SUMMARY:
Obesity interventions in early childhood are recommended as they have been proven to be more effective than interventions later in life. The overall aim of this study is to assess the effectiveness, feasibility, and acceptance of an overweight and obesity intervention in socially disadvantaged families. Participants will be families with children aged 2-6 years (n = 300) with overweight or obesity and will be recruited from three sites: Stockholm, Sweden (n = 100); Timisoara, Romania (n = 100); and Mallorca, Spain (n = 100).

DETAILED DESCRIPTION:
The proposed randomized controlled trial has five specific aims:

Specific Aim 1: To determine the effectiveness of a 10 week parent-only group support program focusing on evidence-based parenting practices followed by a mobile health (mHealth) component for 6-months (n = 150) compared to standard care (n = 150) for overweight and obesity in pre-school children (change in BMI z-scores after 9 months primary outcome).

Specific Aim 2: To determine if the intervention can improve body composition (waist circumference), child eating behaviour, physical activity, and parental feeding practices in comparison to the control group.

Specific Aim 3: To assess reversibility of the molecular signatures of obesity following the intervention through epigenetic markers in white blood cells (methylation) and analyzing the role of the gut hormones.

Specific Aim 4: To assess and validate child food intake with metabolic markers in urine.

Specific Aim 5: To evaluate the feasibility of recruitment (facilitators and barriers), attrition and acceptability, as well as patient and caregiver satisfaction to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 6 year old children with overweight or obesity according to international cut-offs.
* Children who have no other underlying medical condition(s).
* Parent(s) who have the ability to communicate in Swedish (for the Swedish part), Romanian (for the Romanian part), and Spanish (for the Spanish part).

Exclusion Criteria:

* Parent(s) not owning a smartphone compatible with the MINISTOP app.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) z-score. | Baseline, 10 weeks, 9 months, 15 months, 21 months
  It is the most commonly used indicator of changes in weight status in pediatric obesity studies and enable comparison between other studies. The children's weight and height will be measured using standardized procedures and BMI z-scores will be derived from Swedish age and gender specific reference values.

SECONDARY OUTCOMES:
Waist circumference | Baseline, 10 weeks, 9 months, 15 months, 21 months
  Measured at the mid-point between the lower rib and iliac crest.
Eating behaviour | Baseline, 9 months, 15 months, 21 months
  Measured using the Child Eating Behaviour Questionnaire (CEBQ). It includes 35 items on eating styles comprising eight factors related to obesity risk. Parents rate each behavior on a five-point Likert scale. It is a 5-point response scale (''never, rarely, sometimes, mostly, always'' for Items 1-13, and ''disagree, slightly disagree, neutral, slightly agree, agree'' for items 14-49). Mean scores for each subscale will be calculated.
Parenting behaviour | Baseline, 9 months, 15 months, 21 months
  Measured using the Comprehensive Feeding Practices Questionnaire (CFPQ). The CFPQ is a parent-report instrument, designed to measure feeding practices of parents of 2-to-8- year-old children. It contains 49 items comprising 12 factors: 'Encourage Balance and Variety', 'Environment', 'Involvement', 'Modeling', 'Monitoring', 'Teaching about Nutrition', 'Emotion Regulation', 'Food as Reward', 'Pressure', 'Child Control', 'Restriction for Health' and 'Restriction for Weight Control'.
Physical activity and sedentary behaviour | Baseline, 9 months
  Assessed over 7 consecutive days using the ActiGraph wGT3x-BT accelerometer. Children will wear the ActiGraph on the non-dominant wrist 24hrs per day. Parents/caregivers will record when the device has been taken on and off and the activities performed during that time as well as when the child went to bed and woke up. The recorded movements will be used to estimate time in various activity levels (e.g., sedentary behavior, light physical activity etc.) by means of cut-offs.
Food intake | Baseline, 9 months
  First void urinary sample from the child will be collected to assess child food intake. Urine samples will be assessed by proton nuclear magnetic resonance (1H-NMR) spectroscopy. Diet-discriminatory metabolites will be identified so that urine metabolite models can be developed and validated against 24 hour recall data and a food diary for children that attend preschool.
Epigenetic and metabolic markers | Baseline, 9 months
  Fasting blood samples will be collected to assess reversibility of metabolic markers through epigenetic markers and the role of gut hormones. The epigenetic analysis will be carried out in white blood cells, which will required DNA extraction, bisulphite transformation and analysis with specific PCRs or other technologies involving hypothesis-driven CpGs. The unit of measurement/criteria will be changes in percentage of methylation (CpGs). These measurements will be related to other measurements, i.e.: metabolomics and anthropometric measurements. With all the measurements (anthropometrical, and biochemical/genomics) the final purpose would be to build a predictive score of changes related to weight status.
Feasibility, attrition, and acceptability of the intervention as assessed using semi-structured interviews with parents and health care professionals | Baseline, 4 months
  In this qualitative assesment using semi-structured interviews we will thoroughly assess facilitators and barriers of recruitment as well as attrition to the intervention and feasibility and acceptability of the care offered. Both parents and health care professionals will be interviewed by trained staff in the research group post intervention. The interviews are recorded and fully transcribed before they are coded and analyzed using thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Nowicka, Principal Investigator — Karolinska Institutet
Locations (3):
- University of Medicine and Pharmacy "Victor Babes", Timișoara, Romania
- University of the Balearic Islands & CIBEROBN, Palma de Mallorca, Spain
- Karolinska Instituet, Huddinge, Sweden

REFERENCES:
- [Derived] Eli K, Neovius C, Nordin K, Brissman M, Ek A. Parents' experiences following conversations about their young child's weight in the primary health care setting: a study within the STOP project. BMC Public Health. 2022 Aug 12;22(1):1540. doi: 10.1186/s12889-022-13803-8. PMID 35962359
- [Derived] Serban CL, Putnoky S, Ek A, Eli K, Nowicka P, Chirita-Emandi A. Making Childhood Obesity a Priority: A Qualitative Study of Healthcare Professionals' Perspectives on Facilitating Communication and Improving Treatment. Front Public Health. 2021 Jul 15;9:652491. doi: 10.3389/fpubh.2021.652491. eCollection 2021. PMID 34336760
- [Derived] Sjunnestrand M, Nordin K, Eli K, Nowicka P, Ek A. Planting a seed - child health care nurses' perceptions of speaking to parents about overweight and obesity: a qualitative study within the STOP project. BMC Public Health. 2019 Nov 9;19(1):1494. doi: 10.1186/s12889-019-7852-4. PMID 31706318
- [Derived] Ek A, Delisle Nystrom C, Chirita-Emandi A, Tur JA, Nordin K, Bouzas C, Argelich E, Martinez JA, Frost G, Garcia-Perez I, Saez M, Paul C, Lof M, Nowicka P. A randomized controlled trial for overweight and obesity in preschoolers: the More and Less Europe study - an intervention within the STOP project. BMC Public Health. 2019 Jul 15;19(1):945. doi: 10.1186/s12889-019-7161-y. PMID 31307412